CLINICAL TRIAL: NCT05238636
Title: The Effect of Anti-reflux Procedures (Stretta, LINX, and Fundoplication) on Physiological Parameters Contributing to Symptom Resolution in Adults With Gastro-oesophageal Reflux at a Single UK Tertiary Centre
Brief Title: Gastro-intestinal Physiology After Anti-Reflux Procedures
Acronym: GASP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: Wingate Institute of Neurogastroenterology (Other)
Responsible Party: Sponsor
Other Study IDs: 2021.0212; 296193 (Other: IRAS)
Record Dates: First submitted 2022-01-20; First posted 2022-02-14 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Gastroesophageal Reflux
Keywords: Stretta; Laparoscopic fundoplication; LINX
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4-6 oesophageal mucosal biopsies will be taken during endoscopy using standard 2.8 millimetre gastroscopy biopsy forceps and placed into formalin solution then stored in a medical freezer at St George's Hospital. They will then be couriered on dry ice to the Wingate Institute of Neurogastroenterology, where they will undergo immunohistochemical analysis, after which they will be disposed of by standard practices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stretta: Patients that have undergone or are to undergo the Stretta procedure
  Interventions: Procedure: Anti-reflux surgery - Stretta procedure or LINX device or laparoscopic fundoplication
- LINX: Patients that have undergone or are to undergo the LINX device
  Interventions: Procedure: Anti-reflux surgery - Stretta procedure or LINX device or laparoscopic fundoplication
- Laparoscopic fundoplication: Patients that have undergone or are to undergo laparoscopic fundoplication.
  Interventions: Procedure: Anti-reflux surgery - Stretta procedure or LINX device or laparoscopic fundoplication

INTERVENTIONS:
Procedure: Anti-reflux surgery - Stretta procedure or LINX device or laparoscopic fundoplication — This is an observational study. Patients will choose which anti-reflux procedure (Stretta, LINX or fundoplication) they undergo with their clinician, as is standard practice, after which they will be offered recruitment to this study, which will perform investigations to assess for changes in physiology and symptoms.

SUMMARY:
Gastro-oesophageal reflux disease (GORD) affects 1 in 4 adults and is a condition where stomach acid leaks back up into the oesophagus (gullet). It can cause an uncomfortable burning feeling in the chest and even lead to problems such as cancer of the oesophagus. Thankfully most people feel better by changing their diet or taking medications, but for others it can be severe, and they may need to consider having surgery to tighten the internal muscles and stop acid leaking back up. The most common operation is the "laparoscopic fundoplication", which is a keyhole procedure where the top of the stomach is wrapped around the lower oesophagus. Alternatively, the "LINX device" is a keyhole procedure where a magnetic bracelet is placed around the lower oesophagus. The "Stretta procedure" is a non-surgical option, where a probe is placed in the mouth to the oesophagus, where heat energy is applied to strengthen the muscles. All three procedures have been shown to be effective at helping people feel better, but less is known about how exactly they do this and there are not many studies that have been done to compare these procedures.

This study will perform tests on adult patients at St George's University Hospitals NHS Foundation Trust before and again 6 months after their surgery (laparoscopic fundoplication, LINX device or Stretta procedure). The tests are safe and are mostly performed in routine care.

The tests will analyse how surgery affects:

* the strength of the oesophagus muscles
* the amount of acid leaking up
* how sensitive the oesophagus is to acid
* symptoms

This should help lead to a better understanding of what changes are important to make people feel better from GORD and help inform treatment decisions with patients in future.

DETAILED DESCRIPTION:
GORD is caused by backflow of stomach contents, including acid and bile into the oesophagus. It can lead to distressing symptoms such as heartburn, regurgitation, and chest pain. It is more common in men, smokers, advanced age, obesity and consumption of fatty foods and alcohol. The mechanism of GORD can be complex and multifactorial. The best appreciated mechanism is reduced pressure of the lower oesophageal sphincter (LOS) or excessive transeient relaxations of the LOS (TLOSR), which allows stomach contents to reflux into the oesophagus. Hiatus hernia can cause GORD by a similar mechanism as the stomach is displaced upwards into the chest due to weakness of the diaphragm muscle.

Laparoscopic fundoplication and LINX are the most commonly performed anti-reflux surgery (ARS) and are procedures designed to increase the tightness of the LOS. The Stretta procedure is a mimimally invasive and non-surgical anti-reflux procedure, first develped in 2000 and has been gaining in popularity and interest. It involves a balloon catheter being introduced via the mouth to the oesophagus, in a sedated or anaesthetised patient. Gastroscopy is performed first to establish the location of the gastro-oesophageal junction (GOJ). The Stretta catheter then deploys four 5.5mm needle electrodes into the mucosa 1cm above the GOJ. Radiofrequency energy is deployed through the needles to achieve a target temperature fo 85°C for 1 minute. The device is then repostioned to target the electrodes on a total of 56 sites in in the lower oesophagus and gastric cardia. The mechanism of action remains poorly understood. It is thought to cause local inflammation and muscular thickening of the LOS, but objective evidence for this is lacking. Studies on Stretta have been small and often retrospective and there is also a paucity of UK data. A systematic review and meta-analysis by Fass et al. in 2017 concluded that Stretta significantly improved quality of life, reduced acid suppressing medication use and reduced oesophageal acid exposure time, but statistical significance was not reached with regards to its effect on LOS pressure; leading to much ongoing debate about its mechanism of action.

Liu et al (2014) performed a small study showing that oesophageal inflammation/erosions were reduced 6 months following Stretta, again justifying that Stretta is an effective treatment for GORD. The main hypotheses in the literatrure for the mechanism of action of Stretta involve increasing LOS basal pressure, reducing transient LOS relaxations (TLOSRs) and reducing oesophageal sensitivity; with no clear consensus. Tam et al (2003), on a study with 20 patients, showed that Stretta reduced TLOSRs, increased basal LOS pressure and reduced oesophageal acid exposure time at 6 months. Arts et al (2012) gave sildenafil, a smooth muscle relaxant, to 22 patients 3 months after Stretta. They found that sildenafil was able to reduce the LOS pressure, suggesting that the improvement in acid exposure was not due to scarring/fibrosis of the LOS and was therefore due to increased muscle tone.

Further evaluation of LOS function is therefore needed to ascertain how Stretta improves symptoms. EndoFLIP is an endoscopic technique using specialised balloon catheter with pressure sensors that can be placed at the gastro-oesophageal junction at the time of gastroscopy to determine the pressure and distensibility of the GOJ. Kwiatek et al (2010) first described its applicability to GORD, showing that in a sample of 20 patients GOJ distensibility was increased two-fold in GORD patients compared controls. More recently, retrospective analysis of nearly 600 patients by Lee et al (2021) showed that GOJ distensibility was again increased in both erosive and non-erosive GORD, compared to healthy controls. The applicability of EndoFLIP following ARS is not yet known. There are only 5 small published studies regarding EndoFLIP after fundoplication, as described in systematic review by Desprez et al (2020), showing that GOJ distensibility was reduced, but methods varied and the correlation with symptomatic outcomes was uncertain. The application of EndoFLIP to GORD and oesophageal disorders is increasingly being appreciated yet there are no published studies looking at EndoFLIP post LINX or Stretta - this project would be the first to do this, as well as further evaluate its use post fundoplication. GOJ distensibility has been shown to be increased in GORD, and it is hypothesised that it will be reduced by Stretta, LINX and fundoplication, and can thus be a useful measure of response to treatment.

Acid perfusion testing (the Bernstein test) is a test of oesophageal sensitivity and is performed by infusing 0.1M hydrochloric acid into the oesophagus via a nasogastric catheter to see if the symptoms of GORD are reproduced. Arts et al (2019) performed the Bernstein test on 13 patients post Stretta and found that oesophageal sensitivity to acid was reduced, suggesting that Stretta made the oesophagus less sensitive to acid. Further evaluation of oesophageal sensitivity to acid post ARS is therefore needed. Another marker for oesophageal sensitivity may be the calcitonin gene related peptide (CRRP), which Xu et al (2013) showed was a marker for afferent sensory nerves in the oesophageal mucosa and was more abundant in those with non-erosive GORD, suggesting its role as a marker of oesophageal sensitivity. CGRP has never been evaluated post ARS - this project would be the first to do this, alongside the Bernstein test.

This study is unique as it will prospectively obtain detailed objective information of oesophageal physiology, using state of the art techniques, pre and post three different ARS, alongside validated symptom assessment, to allow for comparison in efficacy and mechanism of action for symptomatic improvement for Stretta, fundoplication and LINX.

The objective is to obtain detailed information on physiology and GORD symptoms before and 6 month following Stretta, LINX or fundoplication. The investigators will look for changes to explain symptomatic improvement and examine differences between the three ARS procedures.

Outcomes include:

• LOS pressure

* This will be measured with high resolution oesophageal manometry. The investigators will look to see if there is an increase in LOS pressure in each of three ARS and how well this correlates with oesophageal acid exposure and symptom improvement. It is expected that with increased LOS pressure, symptoms of acid reflux will be improved.

  • LOS distensibility
* This will be measured with EndoFLIP. The investigators will look to see if there is a statistically significant difference in LOS distensibility between the three anti-reflux procedures and how well this correlates with oesophageal acid exposure, LOS pressure and symptom improvement. The investigators would expect that with reduced LOS distensibility oesophageal acid exposure will also be reduced. It is expected that fundoplication and LINX to have greater reductions in LOS distensibility compared to Stretta, due to the anatomical disruption of these surgeries.

  • Oesophageal acid exposure
* This will be measured with either 24hr ambulatory pH/impedance nasogastric catheter with symptom association, or with 96hr wireless oesophageal Bravo pH capsule. The investigators will look to see if there is a significant difference in oesophageal acid exposure between the three anti-reflux procedures and if this correlates with symptom improvement. It is expected that with reduced oesophageal acid exposure symptoms will improve.

  • Oesophageal sensitivity to acid
* This will be measured with the Bernstein test. The investigators will look to see whether the three ARS anti-reflux procedures reduce the sensitivity of the oesophagus to acid. It is hypothesised that sensitivity to acid will be most reduced by Stretta, due to the thermal injury caused by the procedure.

  • Gastroscopy
* The investigators will look to characterise the endoscopic appearances of the oesophagus pre and post anti-reflux procedure, including the macroscopic presence of oesophagitis and hiatus hernia. In patients known to have erosive reflux oesophagitis, it is hypothesised this to be improved following their anti-reflux procedure.

  • Oesophageal biopsies
* During gastroscopy, oesophageal biopsies will be taken for immunohistochemical analysis for calcitonin gene-related peptide (CGRP), which is a marker of afferent sensory neurons. Previous studies have shown this to be related to oesophageal sensitivity and that it is more superficial in the oesophageal mucosa in patients with oesophageal hypersensitivity. The investigators will look to see whether anti-reflux procedures affect the presence and location of CGRP, which may contribute to improvement in symptoms. It is hypothesised that this will be reduced by Stretta due to the thermal injury but unchanged by fundoplication and LINX.

  • Symptoms
* This will be objectively assessed with validated symptom questionnaires - Hull Airway Reflux Questionnaire (HARQ), Reflux Symptom Index (RSI), Hospital Odynophagia and Dysphagia Questionnaire (HODQ), Reflux Disease Questionnaire (RDQ), Epworth Sleepiness Scale, and GERD-HRQL. The investigators will look to see if there is a statistically significant improvement in symptoms between the anti-reflux procedures.

  • Use of acid suppressing medications
* The investigators will ask patients if they are requiring acid suppressing medication such as PPI following their anti-reflux procedure. It is expected that PPI use will reduce following their procedure.

The aim is to determine how the Stretta procedure affects the functioning of the oesophagus with physiological testing, and how well it improves reflux symptoms, in comparison to other surgical anti-reflux procedures.

This gap in understanding is important to address. By understanding the mechanism of action of the Stretta procedure, in comparison to fundoplication and LINX, the investigators will better appreciate which patients are most likely to benefit from being offered it. It will also further knowledge of the pathophysiology of GORD and which factors are important for symptom resolution, which will in turn better inform decisions with patients with regards to their symptoms and ARS, and may lead to the development of other more specialised minimally invasive anti-reflux procedures in future.

ELIGIBILITY:
Inclusion Criteria:

* Patient under the care of St George's University Hospital NHS Foundation Trust, London
* Decision to specifically undergo Stretta procedure, laparoscopic fundoplication or LINX device (N.B. this study will have no involvement in that decision or choice of procedure)
* Symptoms compatible with GORD, e.g. heartburn, regurgitation, chest pain
* Physiological evidence of GORD, e.g. endoscopy, HRM, pH studies
* Male or Female
* Age 18 to 90

Exclusion Criteria:

* Patients < 18 years old or >90 years old
* Patients with significant medical co-morbidities
* Patients unable to provide consent for study participation
* Patients unable to easily attend hospital for the physiological tests
* Patients who have had complications from their anti-reflux procedure
* Patients who have previously undergone oesophageal surgery

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients at St George's University Hospitals NHS Foundation Trust, who have been listed for Stretta procedure, LINX device or laparoscopic fundoplication for GORD.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Lower oesophageal sphincter (LOS) pressure | Before and again 6 months after anti-reflux surgery
  Measured in mm Hg with high resolution oesophageal manometry
Gastro-oesophageal junction (GOJ) distensibility index | Before and again 6 months after anti-reflux surgery
  EndoFLIP will be performed to calculate teh GOJ-distensibility index (DI) by dividing the median GOJ-midline cross-sectional area (CSA) by the median intra-balloon pressure over the duration of the 60mL distension, in mm2/mmHg.
Oesophageal acid exposure | Before and again 6 months after anti-reflux surgery
  24hour ambulatory pH monitoring and 96hour BRAVO capsule placement used to calculate % of time lower oesophageal pH is < 4 (normal is <6%)
Oesophageal sensitivity to acid | Before and again 6 months after anti-reflux surgery
  Measured with Bernstein test (0.1M hydrochloric acid oesophageal perfusion) as time (min) to reproduce symptoms of GORD
Oesophageal biopsies | Before and again 6 months after anti-reflux surgery
  Immunohistochemistry to measure the density of calcitonic related gene peptide (CRGP)
Symptoms | Before and again 6 months after anti-reflux surgery
  Hull Airway Reflux Questionnaire (HARQ), Reflux Symptom Index (RSI), Hospital Odynophagia and Dysphagia Questionnaire (HODQ), Reflux Disease Questionnaire (RDQ), Epworth Sleepiness Scale, and GERD-HRQL symptom questionnaires to grade symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jamal Hayat, Study Director — St George's University Hospitals NHS Foundation Trust; Joseph Cooney, Principal Investigator — St George's University Hospitals NHS Foundation Trust
Locations (1):
- St Georges University Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frazzoni M, Piccoli M, Conigliaro R, Frazzoni L, Melotti G. Laparoscopic fundoplication for gastroesophageal reflux disease. World J Gastroenterol. 2014 Oct 21;20(39):14272-9. doi: 10.3748/wjg.v20.i39.14272. PMID 25339814
- [Background] Schizas D, Mastoraki A, Papoutsi E, Giannakoulis VG, Kanavidis P, Tsilimigras D, Ntourakis D, Lyros O, Liakakos T, Moris D. LINX(R) reflux management system to bridge the "treatment gap" in gastroesophageal reflux disease: A systematic review of 35 studies. World J Clin Cases. 2020 Jan 26;8(2):294-305. doi: 10.12998/wjcc.v8.i2.294. PMID 32047777
- [Background] Triadafilopoulos G. Stretta: a valuable endoscopic treatment modality for gastroesophageal reflux disease. World J Gastroenterol. 2014 Jun 28;20(24):7730-8. doi: 10.3748/wjg.v20.i24.7730. PMID 24976710
- [Background] Trudgill NJ, Sifrim D, Sweis R, Fullard M, Basu K, McCord M, Booth M, Hayman J, Boeckxstaens G, Johnston BT, Ager N, De Caestecker J. British Society of Gastroenterology guidelines for oesophageal manometry and oesophageal reflux monitoring. Gut. 2019 Oct;68(10):1731-1750. doi: 10.1136/gutjnl-2018-318115. Epub 2019 Jul 31. PMID 31366456
- [Background] Desprez C, Roman S, Leroi AM, Gourcerol G. The use of impedance planimetry (Endoscopic Functional Lumen Imaging Probe, EndoFLIP(R) ) in the gastrointestinal tract: A systematic review. Neurogastroenterol Motil. 2020 Sep;32(9):e13980. doi: 10.1111/nmo.13980. PMID 32856765
- [Background] BERNSTEIN LM, BAKER LA. A clinical test for esophagitis. Gastroenterology. 1958 May;34(5):760-81. No abstract available. PMID 13538145
- [Background] Sawada A, Lei WY, Zhang M, Lee C, Ustaoglu A, Chen CL, Sifrim D. Esophageal mucosal sensory nerves and potential mechanoreceptors in patients with ineffective esophageal motility. Neurogastroenterol Motil. 2022 Feb;34(2):e14205. doi: 10.1111/nmo.14205. Epub 2021 Jun 21. PMID 34152070
- [Background] Lawenko RM, Lee YY. Evaluation of Gastroesophageal Reflux Disease Using the Bravo Capsule pH System. J Neurogastroenterol Motil. 2016 Jan 31;22(1):25-30. doi: 10.5056/jnm15151. PMID 26717929
- [Background] Chan Y, Ching JY, Cheung CM, Tsoi KK, Polder-Verkiel S, Pang SH, Quan WL, Kee KM, Chan FK, Sung JJ, Wu JC. Development and validation of a disease-specific quality of life questionnaire for gastro-oesophageal reflux disease: the GERD-QOL questionnaire. Aliment Pharmacol Ther. 2010 Feb 1;31(3):452-60. doi: 10.1111/j.1365-2036.2009.04187.x. Epub 2009 Oct 31. PMID 19878152